CLINICAL TRIAL: NCT05718141
Title: An Online Wellness Intervention for University Students: Investigating the Efficacy of The Common Elements Toolbox in the UK
Brief Title: An Online Wellness Intervention for University Students
Acronym: COMET-GB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Reading (Other); King's College London (Other); University of Roehampton (Other); University of Pennsylvania (Other); Newcastle University (Other)
Responsible Party: Principal Investigator, Dr Maria Loades, Clinical Psychologist, Reader in Clinical Psychology, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMET-GB
Record Dates: First submitted 2022-12-19; First posted 2023-02-08 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Mental Health Wellness 1
Keywords: university students; single session intervention; online; self-help; mental well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Parallel groups (1:1 allocation) Randomised controlled trial (RCT) design, with a waiting list control group who will have the opportunity to access the intervention at the end of the follow-up period (i.e. 4 weeks after randomisation).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: COMET-GB (Experimental): Online single session intervention via qualtrics (any internet connected device) based on cognitive and behavioural principles.
  Interventions: Other: COMET-GB
- Waiting List Control (No Intervention): Participants in the control arm will be provided with information about sources of wellbeing support they can access and will also be asked to fill out additional questionnaires at baseline, which will act as a control for time spent completing online activities. These measures are a Symptom Importance Rating Questionnaire, the Chalder Fatigue Questionnaire [32], Pittsburgh Sleep Quality Index [33], Snaith-Hamilton Pleasure Scale [34], Fatigue Associated with Depression Scale [35]. These will not be completed by the intervention group nor reported as main outcomes on the RCT itself, but will be used in separate observational projects.

INTERVENTIONS:
Other: COMET-GB — Online self-guided single session intervention - comprised of 4 modules based on the core principles of CBT, combined with principles from positive psychology. Each module includes short reading exercises, informational videos, and writing exercises.
  * Cognitive Restructuring (labelled "Flexible Thinking")
  * Behavioural Activation (labelled "Positive Activities")
  * Gratitude
  * Self-Compassion
  The initial intervention modules and assessment will take participants approximately 60-75 minutes to complete (15-20 minutes for the assessment measures only).
  Arms: Intervention: COMET-GB

SUMMARY:
The investigators want to understand the impact of a short online single session programme to improve well-being. Therefore, the investigators are investigating a self-help mental health intervention composed of four distinct modules, all designed to be completed within a single, 60-minute online session.Any university student in the UK can take part. Participants are randomly allocated to either:

1. Complete the COMET programme (lasting about 60 minutes) and to practice the skills learned over the next few weeks. Participants are asked to fill out online questionnaires (10-15 minutes) at two points in the future: two weeks from baseline, and four weeks from baseline.

   Or
2. Complete a few extra online questionnaires (lasting about 20-30 minutes), and fill out brief questionnaires (10-15 minutes) two weeks and four weeks later. After filling out the questionnaires in four weeks time, participants will then have the opportunity to complete the COMET programme (lasting about 60 minutes).

DETAILED DESCRIPTION:
The study will use a randomised controlled trial (RCT) design, with a waiting list control (treatment as usual) group who will have the opportunity to access the intervention 4 weeks after randomisation. The intervention is digital and delivered online via Qualtrics. Participants will answer questions before completing the intervention, and at 2-week and 4-week follow-up. The single session intervention is expected to take < 1 hour to complete, with the research study components taking <20 minutes to complete.

ELIGIBILITY:
The target population for this study are undergraduate and postgraduate students at UK universities. To be eligible to participate, an individual must be: (i) a registered undergraduate or postgraduate student at a university in the UK; and (ii) able to access the internet. Those who cannot access the internet will not be eligible, and neither will those who are under 16 years of age.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Well-being | 4 weeks post randomisation
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) - has 14 items that captures participants feelings and thoughts that best describe their experience over the previous 2 weeks using a scale from 1 to 5. Higher scores indicate better wellbeing.

SECONDARY OUTCOMES:
Depressive symptoms | 2 weeks, 4 weeks post randomisation
  Patient Health Questionnaire-9 (PHQ-9), a commonly used measure for depressive symptoms. The PHQ-9 has 9 items which capture the frequency of depressive symptoms over the preceding two weeks using a scale from 0-3. A score of 0-4 indicates no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15- 19 indicates moderately severe depression and 20-24 indicates severe depression. The PHQ-9 has a sensitivity and specificity of 88% for detecting clinical depression.
Anxiety symptoms | 2 weeks, 4 weeks post randomisation
  General Anxiety Disorder 7-item Checklist (GAD-7), a commonly used measure for symptoms of anxiety. The GAD-7 has 7 items which capture the frequency of anxious symptoms over the preceding two weeks using a scale from 0-3. A score of 0-4 indicates no anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety and ≥15 indicates severe anxiety. The GAD-7 has a sensitivity and specificity of 89% and 82% respectively.
Positive and negative affect | 2 weeks, 4 weeks post randomisation
  Positive and Negative Affect Schedule (PANAS), a commonly used measure of positive and negative affect. The PANAS has 20 items that captures participants feelings of positive and negative affect over the past week using a scale from 1 to 5.
Well-being | 2 weeks post randomisation
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS), a commonly used measure of well-being. The WEMWBS has 14 items that captures participants feelings and thoughts that best describe their experience over the previous 2 weeks using a scale from 1 to 5. Higher scores indicate better wellbeing.

OTHER OUTCOMES:
Acceptability (intervention arm only) | Immediately post intervention
  Acceptability of Interventions Measure (AIM)
Appropriateness (intervention arm only) | Immediately post intervention
  Intervention Appropriateness Measure (IAM)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Banes, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2024 - ongoing
Access Criteria: Proof of researcher status.

REFERENCES:
- [Derived] Lambert J, Loades M, Marshall N, Higson-Sweeney N, Chan S, Mahmud A, Pile V, Maity A, Adam H, Sung B, Luximon M, MacLennan K, Berry C, Chadwick P. Investigating the Efficacy of the Web-Based Common Elements Toolbox (COMET) Single-Session Interventions in Improving UK University Student Well-Being: Randomized Controlled Trial. J Med Internet Res. 2025 Jan 31;27:e58164. doi: 10.2196/58164. PMID 39888663